CLINICAL TRIAL: NCT00288145
Title: Statewide Partnerships for Worksite Weight Management
Brief Title: Statewide (Rhode Island and Neighboring States) Partnerships for Worksite Weight Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kim Gans, Director, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R18DK071946 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Overweight; Obesity
Keywords: worksite; weight gain prevention (among adults); obesity (among adults); physical activity; nutrition
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T (Active Comparator): Treatment arm comprises one worksite in a matched site pair; one site assigned to treatment, the other site assigned to comparison. Treatment site worksite-based health promotion activities such as self-directed campaigns, lectures, small group programs, online programs, environment interventions (food service and physical)--all with focus on nutrition, physical activity and/or weight management.
  Interventions: Behavioral: WOW, Working On Wellness weight management

INTERVENTIONS:
Behavioral: WOW, Working On Wellness weight management — Treatment site, worksite-based health promotion activities such as self-directed campaigns, lectures, small group programs, online programs, environment interventions (food service and physical)--all with focus on nutrition, physical activity and/or weight management.

SUMMARY:
The project is designed to test the effectiveness of a multilevel worksite wellness program, based in Rhode Island and nearby neighboring states to impact employee weight, dietary intake and physical activity, compared to an attention placebo condition.

DETAILED DESCRIPTION:
Accomplishment of the specific aim will be determined by a two group randomized effectiveness study (Treatment vs. Comparison) utilizing 24 RI worksites with randomization by site. The specific impact and outcome evaluation measures (BMI, DHQ-FFQ, and 7-day PAR) will be collected at Baseline, 12, and 24 months on a longitudinal cohort selected at random from the employee lists of each participating worksite. Extensive process evaluation and a mediating variable framework are also included to identify the mechanisms in successful change at both the worksite and individual level, which will maximize the potential for dissemination and generalization of the intervention as well as advance theory and improve intervention practice and policy.

Primary outcome measure will be weight (BMI).

ELIGIBILITY:
Inclusion Criteria:

Worksite

* worksite located in Rhode Island or neighboring state
* has food service on site
* approximately 200 - 500 employees
* low rate of employee turnover

Exclusion Criteria:

* worksites outside New England

Cohort participants:

* permanent employee, who works 20 or more hours on site
* speaks/reads some English at level to complete survey eval items
* able to walk at a brisk pace

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2006-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Weight (BMI) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Gans, PhD MPH LDN, Principal Investigator — Brown University, Institute for Community Health Promotion
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Background] Proper KI, Koning M, van der Beek AJ, Hildebrandt VH, Bosscher RJ, van Mechelen W. The effectiveness of worksite physical activity programs on physical activity, physical fitness, and health. Clin J Sport Med. 2003 Mar;13(2):106-17. doi: 10.1097/00042752-200303000-00008. PMID 12629429
- [Background] Hallam JS, Petosa R. The long-term impact of a four-session work-site intervention on selected social cognitive theory variables linked to adult exercise adherence. Health Educ Behav. 2004 Feb;31(1):88-100. doi: 10.1177/1090198103259164. PMID 14768660
- See also: American Council on Fitness and Nutrition website — http://www.acfn.org/